CLINICAL TRIAL: NCT00707291
Title: Characterization of the Edge of Soft Contact Lens and Its Interaction With Ocular Surface
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Jianhua (Jay) Wang, MD, PhD, Associate Professor, University of Miami
Other Study IDs: UMOCT9010_Vis_Edge
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: contact lens; normal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to look at contact lens on the eye and its interaction with the eye during wearing.

DETAILED DESCRIPTION:
The goal of this study is to characterize the edge of contact lenses and its interaction with ocular surface.

ELIGIBILITY:
Inclusion Criteria:

* self reported normal subjects

Exclusion Criteria:

* any ocular diseases/conditions
* will not wear contact lenses

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
difference characteristics with different contact lenses and different interactions with the eye | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Insititute, Miami, Florida, United States